CLINICAL TRIAL: NCT02030067
Title: A Phase 1, Open-Label, Dose-Ranging, Safety and Pharmacokinetic Study to Determine the Maximum Tolerated Dose of RX-3117 Administered Orally as a Single-Agent to Subjects With Advanced Malignancies
Brief Title: Dose-Finding and Safety Study for Oral Single-Agent to Treat Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RX-3117-P1-01
Record Dates: First submitted 2013-12-24; First posted 2014-01-08 (Estimated); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumor; Metastatic Bladder Cancer
Keywords: oncology; tumor; metastatic; bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — fluorocyclopentenylcytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RX-3117 (Experimental): All subjects will receive RX-3117.
  Interventions: Drug: RX-3117

INTERVENTIONS:
Drug: RX-3117

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of RX-3117 in subjects with advanced or metastatic solid tumors (Phase 1). The purpose of the Phase 2 portion is to estimate anti-tumor activity in subjects with advanced malignancies (relapsed or refractory pancreatic or advanced bladder cancer).

DETAILED DESCRIPTION:
This is a dose-finding, open-label, single agent study of RX-3117. Once the maximum tolerated dose is identified additional subjects will be treated in a dose expansion followed by a 2-stage Phase 2 study. Subjects will be treated for up to 8 cycles of therapy. A cycle will be 4 weeks. RX-3117 dosing will be 3 times each week for 3 weeks follow by 1 week off treatment. All subjects will be followed for at least 30 days after the last dose of RX-3117.

ELIGIBILITY:
Inclusion Criteria:

* Males or females who are 18 years or older
* Able to swallow capsules
* Histological or cytological evidence of confirmed metastatic pancreatic or advanced bladder cancer
* Able to discontinue all anticancer therapies 2 weeks prior to study start
* Measurable or evaluable disease using Response Evaluation Criteria in Solid Tumors
* Life expectancy of at least 3 months
* ECOG performance status of 0 or 1
* Provide written informed consent

Exclusion Criteria:

* Primary brain tumors or clinical evidence of active brain metastasis
* Systemic corticosteroid use within 7 days before planned start of study therapy
* Active infection requiring parenteral or oral antibiotics within 2 weeks before planned start of study therapy
* Uncontrolled diabetes as assessed by the investigator
* Prior or current history of hepatitis B, hepatitis C or human immunodeficiency virus
* History of bone marrow of solid organ transplantation
* History of congestive heart failure, arrhythmias, acute coronary syndrome or torsades de pointes
* Any other medical, psychiatric, or social condition, which in the opinion of the investigator, would preclude participation in the study, pose an undue medical hazard, interfere with the conduct of the study, or interfere with interpretation of the study results
* Known hypersensitivity to gemcitabine, azacytidine or cytosine arabinoside
* Pregnant, planning a pregnancy or breast feeding during the study
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2013-12; Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ely Benaim, MD, Study Director — Rexahn Pharmaceuticals, Inc.
Locations (12):
- United States (12):
  - Rexahn Site, Birmingham, Alabama
  - Rexahn Site, Tucson, Arizona
  - Rexahn Site, Duarte, California
  - Rexahn Site, Miami, Florida
  - Rexahn Site, Miami Lakes, Florida
  - Rexahn Site, Skokie, Illinois
  - Rexahn Site, St Louis, Missouri
  - Rexahn Site, Las Vegas, Nevada
  - Rexahn Site, New York, New York
  - Rexahn Site, San Antonio, Texas
  - Rexahn Site, Salt Lake City, Utah
  - Rexahn Site, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients enrolled in the Phase 2 portion of the study discontinued prior to dosing. Therefore 124 patients started the study rather than 127 patients as listed in the protocol section.
Groups:
- RX-3117 30 mg, 3 Times/Week: Subjects will receive 30 mg RX-3117, 3 times/week
- RX-3117 60 mg, 3 Times/Week: Subjects will receive 60 mg RX-3117 3 times/week
- RX-3117 100 mg, 3 Times/Week: Subjects will receive 100 mg RX-3117 3 times/week
- RX-3117 150 mg, 3 Times/Week: Subjects will receive 150 mg RX-3117, 3 times/week
- RX-3117 200 mg, 3 Times/Week: Subjects will receive 200 mg of RX-3117, 3 times/week
- RX-3117 500 mg, 3 Times/Week: Subjects will receive 500 mg RX-3117, 3 times/week
- RX-3117 1000 mg, 3 Times/Week: Subjects received 1000 mg RX-3117, 3 times/week
- RX 3117 1500 mg, 3 Times/Week: Subjects received 1500 mg RX-3117, 3 times/week
- RX-3117 2000 mg, 3 Times/Week: Subjects received 2000 mg RX-3117, 3 times/week
- RX-3117 500 mg, 5 Times/Week: Subjects receivved 500 mg RX-3117, 5 times/week
- RX-3117 700 mg, 5 Times/Week: Subjects received 700 mg RX-3117, 5 times/week
- RX-3117 500 mg, 7 Times/Week: Subjects received 500 mg RX-3117, 7 times/week
- RX-3117 700 mg 5 Times/Week (Phase 2 Portion of Study): Subjects received MTD of 700 mg RX-3117, 5 times/week
Period: Overall Study
Arm/Group | RX-3117 30 mg, 3 Times/Week | RX-3117 60 mg, 3 Times/Week | RX-3117 100 mg, 3 Times/Week | RX-3117 150 mg, 3 Times/Week | RX-3117 200 mg, 3 Times/Week | RX-3117 500 mg, 3 Times/Week | RX-3117 1000 mg, 3 Times/Week | RX 3117 1500 mg, 3 Times/Week | RX-3117 2000 mg, 3 Times/Week | RX-3117 500 mg, 5 Times/Week | RX-3117 700 mg, 5 Times/Week | RX-3117 500 mg, 7 Times/Week | RX-3117 700 mg 5 Times/Week (Phase 2 Portion of Study)
Started | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 11 | 3 | 80
Completed | 0 (only 1 patient in phase 1 completed; 0 patients in phase 2 completed) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 2 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 11 | 3 | 80
Not completed — Disease Progression | 1 | 1 | 2 | 2 | 3 | 2 | 3 | 3 | 4 | 3 | 7 | 2 | 59
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 6
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — other reasons | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- RX-3117 30 mg 3 Times/Week: Patient received 30 mg RX-3117 3 times/week
- RX-3117 60 mg 3 Times/Week: Patient received 60 mg RX-3117 3 times/week
- RX-3117 100 mg 3 Times/Week: Patients received 100 mg RX-3117 3 times/week
- RX-3117 150 mg 3 Times/Week: Patients received 150 mg RX-3117 3 times/week
- RX-3117 200 mg 3 Times/Week: Patients received 200 mg RX-3117 3 times/week
- RX-3117 500 mg 3 Times/Week: Patients received 500 mg RX-3117 3 times/week
- RX-3117 1000 mg 3 Times/Week: Patients received 1000 mg RX-3117 3 times/week
- RX-3117 1500 mg 3 Times/Week: Patients received 1500 mg RX-3117 3 times/week
- RX-3117 2000 mg 3 Times/Week: Patients received 2000 mg RX-3117 3 times/week
- RX-3117 500 mg 5 Times/Week: Patients received 500 mg RX-3117 5 times/week
- RX-3117 700 mg 5 Times/Week; RX-3117 700 mg 5 Times/Week (Phase 2): Patients received 700 mg RX-3117 5 times/week
- RX-3117 500 mg 7 Times/Week: Patients received RX-3117 500 mg 7 Times/Week
- Total: Total of all reporting groups
Arm/Group | RX-3117 30 mg 3 Times/Week | RX-3117 60 mg 3 Times/Week | RX-3117 100 mg 3 Times/Week | RX-3117 150 mg 3 Times/Week | RX-3117 200 mg 3 Times/Week | RX-3117 500 mg 3 Times/Week | RX-3117 1000 mg 3 Times/Week | RX-3117 1500 mg 3 Times/Week | RX-3117 2000 mg 3 Times/Week | RX-3117 500 mg 5 Times/Week | RX-3117 700 mg 5 Times/Week | RX-3117 500 mg 7 Times/Week | RX-3117 700 mg 5 Times/Week (Phase 2) | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 11 | 3 | 80 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (0) | 66.0 (0) | 65.3 (5.86) | 67.0 (4.58) | 68.0 (6.24) | 53.7 (7.57) | 54.3 (4.16) | 63.3 (16.50) | 61.0 (13.30) | 62.0 (13.08) | 58.0 (10.87) | 67.0 (6.56) | 67.6 (9.11) | 65.37 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2 | 2 | 2 | 3 | 1 | 4 | 2 | 8 | 3 | 34 | 63
  Male | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 3 | 2 | 1 | 3 | 0 | 46 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 3 | 1 | 5 | 1 | 14 | 31
  Not Hispanic or Latino | 1 | 0 | 2 | 2 | 2 | 2 | 1 | 4 | 3 | 2 | 6 | 2 | 63 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 8 | 10
  White | 1 | 1 | 3 | 3 | 3 | 1 | 1 | 3 | 5 | 3 | 9 | 2 | 64 | 99
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety Profile Characterized by # of Subjects With Dose-limiting Toxicities (DLTs) in Phase 1
Description: Number of subjects participating in Phase 1 that experienced a DLT during the first cycle of treatment (28 days)
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 30 mg, 3 Times/Week | RX-3117 60 mg, 3 Times/Week | RX-3117 100 mg, 3 Times/Week | RX-3117 150 mg, 3 Times/Week | RX-3117 200 mg, 3 Times/Week | RX-3117 500 mg, 3 Times/Week | RX-3117 1000 mg, 3 Times/Week | RX 3117 1500 mg, 3 Times/Week | RX-3117 2000 mg, 3 Times/Week | RX-3117 500 mg, 5 Times/Week | RX-3117 700 mg, 5 Times/Week | RX-3117 500 mg, 7 Times/Week
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 11 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2

2. Primary Outcome: Overall Safety Profile Characterized by Number of Subjects Experiencing Serious Adverse Events in Phase 1
Description: Number of subjects participating in Phase 1 that experience any SAEs
Time Frame: through study completion, up to 224 days (8 cycles of treatment)
Population: Population includes those subjects participating in the dose escalation phase of the study (Phase 1)
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 30 mg, 3 Times/Week | RX-3117 60 mg, 3 Times/Week | RX-3117 100 mg, 3 Times/Week | RX-3117 150 mg, 3 Times/Week | RX-3117 200 mg, 3 Times/Week | RX-3117 500 mg, 3 Times/Week | RX-3117 1000 mg, 3 Times/Week | RX 3117 1500 mg, 3 Times/Week | RX-3117 2000 mg, 3 Times/Week | RX-3117 500 mg, 5 Times/Week | RX-3117 700 mg, 5 Times/Week | RX-3117 500 mg, 7 Times/Week
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 11 | 3
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 5 | 1

3. Primary Outcome: Overall Safety Profile Characterized by the Number of Subjects That Discontinue Study Treatment - Phase 1
Description: Number of subjects participating in Phase 1 of study that discontinued study treatment due to a treatment emergent adverse event.
Time Frame: through study completion, up to 224 days (8 cycles of treatment)
Population: Population includes subjects in the dose escalation phase of the study (Phase 1)
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 30 mg, 3 Times/Week | RX-3117 60 mg, 3 Times/Week | RX-3117 100 mg, 3 Times/Week | RX-3117 150 mg, 3 Times/Week | RX-3117 200 mg, 3 Times/Week | RX-3117 500 mg, 3 Times/Week | RX-3117 1000 mg, 3 Times/Week | RX 3117 1500 mg, 3 Times/Week | RX-3117 2000 mg, 3 Times/Week | RX-3117 500 mg, 5 Times/Week | RX-3117 700 mg, 5 Times/Week | RX-3117 500 mg, 7 Times/Week
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 11 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

4. Primary Outcome: Overall Safety Profile Characterized by Number of Subjects Experiencing a Treatment Emergent Adverse Event- Phase 1
Description: Number of subjects that experience any treatment-related adverse event.
Time Frame: through study completion, up to 224 days (8 cycles of treatment)
Population: Population includes subjects participating in the dose escalation phase of the study (Phase 1)
Measure: Count of Participants; unit: Participants
Arm/Group | RX-3117 30 mg, 3 Times/Week | RX-3117 60 mg, 3 Times/Week | RX-3117 100 mg, 3 Times/Week | RX-3117 150 mg, 3 Times/Week | RX-3117 200 mg, 3 Times/Week | RX-3117 500 mg, 3 Times/Week | RX-3117 1000 mg, 3 Times/Week | RX 3117 1500 mg, 3 Times/Week | RX-3117 2000 mg, 3 Times/Week | RX-3117 500 mg, 5 Times/Week | RX-3117 700 mg, 5 Times/Week | RX-3117 500 mg, 7 Times/Week
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 11 | 3
Participants | 0 | 1 | 2 | 3 | 3 | 0 | 2 | 3 | 6 | 3 | 9 | 3

5. Primary Outcome: Progression Free Survival (Phase 2)
Description: Progression Free Survival in Phase 2 of the study for pancreatic and bladder cancer subjects.
Time Frame: 4 months
Population: Patients participating in Phase 2 of the study, which included 41 pancreatic cancer and 31 bladder cancer patients
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | RX-3117 700 mg 5 Times/Week (Phase 2 Portion of Study)
Number analyzed (Participants) | 72
weeks
  Pancreatic cancer patients: number analyzed (Participants) | 41
  Pancreatic cancer patients | 4.7 [3.14 to 8.00]
  Bladder cancer patients: number analyzed (Participants) | 31
  Bladder cancer patients | 7.7 [7.14 to 13.00]

6. Secondary Outcome: Area Under the Plasma Concentration Time Curve (AUC) (Phase 1)
Time Frame: Pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 24 and 48 hours after oral administration in Cycle 1 Days 1 and 15
Population: No pharmacokinetic analysis was conducted
Groups:
- RX-3117: All subjects will receive RX-3117.
  RX-3117
Arm/Group | RX-3117
Number analyzed (Participants) | 0

7. Secondary Outcome: Best Overall Response Rate (Phase 2)
Description: Best Overall Response Rate (includes Complete Response, Partial Response, and Stable Disease)
Time Frame: Baseline and at 4, 8, 12, 16 and 32 weeks
Population: Evaluable for Tumor Response Analysis Set (includes Bladder and Pancreatic patients in Phase 2)
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | RX-3117 700 mg 5 Times/Week (Phase 2 Portion of Study)
Number analyzed (Participants) | 72
percentage
  pancreatic subjects: number analyzed (Participants) | 41
  pancreatic subjects | 26.8 [14.2 to 42.9]
  bladder subjects: number analyzed (Participants) | 31
  bladder subjects | 45.2 [27.3 to 64.0]

8. Other Pre Specified Outcome: Biomarker Concentrations in Blood (Phase 1 and Phase 2)
Description: Analysis of biomarker data not conducted. Biomarker samples were not analyzed due to previous sponsor terminating clinical program.
Time Frame: Baseline and 4, 8, 12, 16 and 32 weeks
Population: Analysis of biomarker data not conducted. Biomarker samples were not analyzed due to previous sponsor terminating clinical program.
Arm/Group | RX-3117 30 mg, 3 Times/Week | RX-3117 60 mg, 3 Times/Week | RX-3117 100 mg, 3 Times/Week | RX-3117 150 mg, 3 Times/Week | RX-3117 200 mg, 3 Times/Week | RX-3117 500 mg, 3 Times/Week | RX-3117 1000 mg, 3 Times/Week | RX 3117 1500 mg, 3 Times/Week | RX-3117 2000 mg, 3 Times/Week | RX-3117 500 mg, 5 Times/Week | RX-3117 700 mg, 5 Times/Week | RX-3117 500 mg, 7 Times/Week | RX-3117 700 mg 5 Times/Week (Phase 2 Portion of Study)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 224 days (8 cycles of treatment)
Groups:
- Phase 1 (Dose Escalation) 30 mg 3x/Week: RX-3117 30 mg administered 3 times/week
- Phase 1 (Dose Escalation) 60 mg 3x/Week: RX-3117 60 mg administered 3 times/week
- Phase 1 (Dose Escalation) 100 mg 3x/Week: RX-3117 100 mg administered 3 times/week
- Phase 1 (Dose Escalation) 150 mg 3x/Week: RX-3117 150 mg administered 3 times/week
- Phase 1 (Dose Escalation) 200 mg 3x/Week: RX-3117 200 mg administered 3 times/week
- Phase 1 (Dose Escalation) 500 mg 3x/Week: RX-3117 500 mg administered 3 times/week
- Phase 1 (Dose Escalation) 1000 mg 3x/Week: RX-3117 1000 mg administered 3 times/week
- Phase 1 (Dose Escalation) 1500 mg 3x/Week: RX-3117 1500 mg administered 3 times/week
- Phase 1 (Dose Escalation) 2000 mg 3x/Week: RX-3117 2000 mg administered 3 times/week
- Phase 1 (Dose Escalation) 500 mg 5x/Week: RX-3117 500 mg administered 5 times/week
- Phase 1 (Dose Escalation) 700 mg 5x/Week; Phase 2 700 mg: RX-3117 700 mg administered 5 times/week
- Phase 1 (Dose Escalation) 500 mg 7x/Week: RX-3117 500 mg administered 7 times/week
Arm/Group | Phase 1 (Dose Escalation) 30 mg 3x/Week | Phase 1 (Dose Escalation) 60 mg 3x/Week | Phase 1 (Dose Escalation) 100 mg 3x/Week | Phase 1 (Dose Escalation) 150 mg 3x/Week | Phase 1 (Dose Escalation) 200 mg 3x/Week | Phase 1 (Dose Escalation) 500 mg 3x/Week | Phase 1 (Dose Escalation) 1000 mg 3x/Week | Phase 1 (Dose Escalation) 1500 mg 3x/Week | Phase 1 (Dose Escalation) 2000 mg 3x/Week | Phase 1 (Dose Escalation) 500 mg 5x/Week | Phase 1 (Dose Escalation) 700 mg 5x/Week | Phase 1 (Dose Escalation) 500 mg 7x/Week | Phase 2 700 mg
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/4 | 0/6 | 0/3 | 1/11 | 0/3 | 8/80
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/3 | 0/3 | 0/3 | 0/3 | 1/3 | 0/4 | 2/6 | 2/3 | 5/11 | 1/3 | 29/80
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 3/3 | 3/3 | 0/3 | 3/3 | 4/4 | 6/6 | 3/3 | 11/11 | 3/3 | 78/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Dose Escalation) 30 mg 3x/Week (N=1) | Phase 1 (Dose Escalation) 60 mg 3x/Week (N=1) | Phase 1 (Dose Escalation) 100 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 150 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 200 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 500 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 1000 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 1500 mg 3x/Week (N=4) | Phase 1 (Dose Escalation) 2000 mg 3x/Week (N=6) | Phase 1 (Dose Escalation) 500 mg 5x/Week (N=3) | Phase 1 (Dose Escalation) 700 mg 5x/Week (N=11) | Phase 1 (Dose Escalation) 500 mg 7x/Week (N=3) | Phase 2 700 mg (N=80)
pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
cervical cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Dose Escalation) 30 mg 3x/Week (N=1) | Phase 1 (Dose Escalation) 60 mg 3x/Week (N=1) | Phase 1 (Dose Escalation) 100 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 150 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 200 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 500 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 1000 mg 3x/Week (N=3) | Phase 1 (Dose Escalation) 1500 mg 3x/Week (N=4) | Phase 1 (Dose Escalation) 2000 mg 3x/Week (N=6) | Phase 1 (Dose Escalation) 500 mg 5x/Week (N=3) | Phase 1 (Dose Escalation) 700 mg 5x/Week (N=11) | Phase 1 (Dose Escalation) 500 mg 7x/Week (N=3) | Phase 2 700 mg (N=80)
nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 6 | 3 | 22
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37
vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 2 | 14
abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 23
constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 9
fatigue (General disorders) | 0 | 1 | 2 | 2 | 2 | 0 | 1 | 3 | 4 | 1 | 6 | 1 | 39
oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 9
decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 15
hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 7
hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 2 | 4 | 2 | 38
neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4
arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 7
dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 5
lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 5
leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
white blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT02030067/Prot_SAP_000.pdf